CLINICAL TRIAL: NCT04012190
Title: Severe Infections and the Intestinal Microbiome in Young Infants in Dhaka, Bangladesh: an Observational Cohort Study
Brief Title: SEPSIS Observational Cohort Study in Young Infants in Bangladesh
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Child Health Research Foundation, Bangladesh (Other); Boston University (Other); McGill University (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Daniel Roth, Scientist, The Hospital for Sick Children
Other Study IDs: 1000063899
Record Dates: First submitted 2019-06-19; First posted 2019-07-09 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Severe Infection and Non-injury Death
Keywords: Severe infection; Sepsis; Microbiome; Bangladesh; Young infants
MeSH Terms: conditions — Infections; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Routine specimen collection:
  1. Infant: stool; nasal, skin, oral swabs; blood. Skin swabs, oral swabs and blood will only be collected in a sub-set of participants.
  2. Maternal: stool, vaginal swabs, breast milk. Stool and vaginal swabs will only be collected in a sub-set of mothers.
  3. Stool sample from a sibling closest in age to the participant will be collected from a subset of participants (excluding twin).
  Specimen collection triggered by presence of clinical severe infection (CSI): infant stool, nasal swab, blood, urine; and, skin swabs and cerebrospinal fluid (CSF) at treating physician's discretion.
  Nasal swabs will also be collected from infants with LRTI (fast breathing with at least one of cough, nasal congestion, or runny nose) or in hospitalized infants with diarrhea and/or vomiting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Globally, infectious diseases such as sepsis, meningitis and pneumonia are among the leading causes of neonatal deaths. A recent observational study in South Asia highlighted the contribution of both bacterial and viral infections to the burden of illness in infants <60 days of age; however, there remains a need to quantify the risk of severe infection (SI) among newborns in a Bangladeshi population. In collaboration with researchers in Bangladesh, investigators aim to generate knowledge regarding the incidence and risk factors of SI, including the composition of the intestinal microbiome, in young infants (birth to 60 days of age) in Dhaka, Bangladesh. Data will support the design and implementation of future trials to test the efficacy of novel interventions for the prevention of SI in young infants, to promote optimal growth and development, and to determine effects on other health outcomes in early infancy.

DETAILED DESCRIPTION:
Globally, infectious diseases including sepsis, meningitis, and pneumonia are among the leading causes of neonatal deaths. In 2017, these three conditions were estimated to account for 540,000 newborn deaths worldwide, approximately 21% of all neonatal deaths globally. Previous studies have suggested that South Asia has a relatively high incidence of possible serious bacterial infection (pSBI) in young infants, particularly in areas where neonatal and under-five mortality rates are highest.

A large body of evidence from inpatient neonatal populations, and the recent evidence from the Panigrahi et al. community trial in India, support an important role of intestinal dysbiosis in the pathogenesis of sepsis/SI in young infants. This mechanism may be particularly important in low- and middle-income countries in Africa and South Asia, where low-cost routine interventions to reduce the burden of SI (e.g., probiotics or synbiotics) could have an important impact on the burden of morbidity and mortality in young infants. However, there are limited data regarding the composition of the early postnatal microbiome in the general population of infants (rather than selected groups of preterm or hospitalized newborns) in South Asia and the role of the microbiome in modulating the risk of SI.

This observational study will generate new knowledge about the incidence and risk factors of SI, including the composition of the intestinal microbiome, in young infants (birth to 60 days of age) in Dhaka, Bangladesh. The aims of this study are to:

1. Estimate the incidence of SI in a facility-recruited cohort of Bangladeshi newborns during the first 60 days of life, and examine the sensitivity of the estimates to variations in SI case definitions;
2. Explore the associations between maternal-infant characteristics (e.g., mode of delivery, feeding practices, gestational age, antibiotic exposure) and the risk of SI in the first 60 days of life;
3. Estimate the absolute and relative stool abundances and age at initial colonization of Bifidobacterium longum subspecies (ssp.) infantis (B. infantis), Bifidobacterium longum ssp. longum (B. longum longum), Bifidobacterium breve (B. breve) and all bifidobacteria species combined during the first 60 days of life in Bangladeshi newborns, overall and within sub-groups defined by: mode of delivery, feeding practices, prior or current infant exposure to antibiotics, and whether there is colonization with the specific bacterial species or subspecies;
4. Explore the associations between maternal-infant characteristics (e.g., mode of delivery, feeding practices, gestational age, antibiotic use) and stool abundance (or age at initial colonization) of B. infantis, B. longum longum, and B. breve;
5. Estimate the association between stool abundance of B. infantis and SI in Bangladeshi newborns during the first 60 days of life;
6. Describe the composition, diversity, and stability of the microbiome in Bangladeshi newborns at multiple time-points during the first 60-days of life, and examine how the composition, diversity, and stability varies by mode of delivery and other maternal-infant and household characteristics;
7. In a facility-recruited cohort of Bangladeshi newborns, estimate the incidence proportions and/or incidence rates and/or prevalence of the following clinical outcomes up to 7 days, 28 days, 60 days of life, 3 months, and 6 months of age:

   1. Hospitalization for any reason other than for routine postnatal care
   2. Upper respiratory tract infections (URTI);
   3. Lower respiratory tract infections (LRTI);
   4. Acute or persistent diarrhea;
   5. Significant neurological impairment or disability diagnosed by 6 months of age; and,
   6. All-cause and non-injury-related mortality
8. Describe child anthropometry (length, weight, and head circumference) and standardized anthropometric indices (length-for-age, weight-for age, and weight-for-height, and head circumference-for-age z-scores) up to 60 days of age in a facility-recruited cohort of Bangladeshi newborns;
9. Estimate the cohort accrual rates of eligible newborns at two public maternal-child health care facilities in Dhaka, Bangladesh

Study personnel will conduct active and passive clinical surveillance and routine specimen collection (e.g. stool, nasal, skin and oral swabs etc.). Additional specimen collection may also be triggered in the event of physician-confirmed clinical severe infection, or if infants meet the case definition of LRTI (fast breathing with at least one of the following: cough, nasal congestion, or runny nose) or are hospitalized with diarrhea and/or vomiting.

ELIGIBILITY:
Core Inclusion Criteria:

* Infants up to and including 4 days of age
* Infants delivered at a study hospital
* Orally feeding currently
* Informed consent by parent or guardian
* Intends to maintain residence within the defined catchment areas (upon discharge from hospital) until 60 days of age

Core Exclusion Criteria:

* Birth weight <1500g
* Death or major surgery considered to be highly probable within first week of life
* Major congenital anomaly of the gastrointestinal tract
* Maternal HIV infection and/or history of mother ever receiving anti-retroviral drug(s) for presumed HIV infection
* Current mechanical ventilation and/or cardiac support (e.g., inotropes) and/or administration/prescription of parenteral antibiotics
* Any prenatal or postpartum use of non-dietary probiotic supplement by mother (during current pregnancy)
* Any postnatal administration of non-dietary probiotic or prebiotic supplements to infant
* Enrolment of infant in any other clinical trial involving the administration of probiotics and/or prebiotics
* Resides in the same household as another infant previously enrolled in the study, or any study within the research platform, who is currently <60 days of age; however, twins may all be enrolled simultaneously
* Multiple gestation for which the number of liveborn infants from the same pregnancy exceeds two (i.e., triplets or higher order multiples)

Ages: 0 Days to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy Bangladeshi newborns, delivered at two public hospitals (Maternal and Child Health Training Institute and Mohammadpur Fertility Services and Training Centre), and their mothers in Dhaka, Bangladesh. Newborns will be enrolled between 0 and 4 days postnatal age (n=3,000).
Sampling Method: Non-Probability Sample
Enrollment: 2083 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-10-22 (Actual)

PRIMARY OUTCOMES:
Incidence of severe infection (SI) and/or non-injury death | Up to 60 days of age
  Severe infection is defined as at least one sign of clinical severe infection (CSI) (i.e., poor feeding, lethargy, convulsions, severe chest in-drawing, fever, or hypothermia) documented by a physician and/or physician diagnosis of sepsis or another serious bacterial infection (SBI); and at least one of the following two criteria: 1) physician decision to admit to hospital, administration of at least one dose of a parenteral antibiotic on the day when CSI/sepsis/SBI is first ascertained, and treatment (or physician intention to treat) with parenteral antibiotics for at least 5 days or 2) blood and/or cerebrospinal fluid (CSF) culture positive for a pathogenic bacterial or fungal organism.
  Non-injury death refers to death due to any cause except death that was directly caused by physical trauma (medically certified cause of death and/or verbal autopsy).
Absolute abundance of Bifidobacterium infantis, Bifidobacterium longum longum and Bifidobacterium breve in stool | Up to 60 days of age
  Absolute abundance (AA) of specific bacteria in stool will be expressed as the log number of cells of a particular bacterial species or subspecies per gram (g) of stool, as detected by quantitative polymerase chair reaction (qPCR). If a direct cell count is unfeasible, AA will be expressed as log colony forming units of a particular bacterial species or subspecies per gram of stool.
Relative abundance of Bifidobacterium infantis, Bifidobacterium longum longum and Bifidobacterium breve in stool | Up to 60 days of age
  Relative abundance (RA) will be expressed as the number of gene copies from a particular genus/species/sub-species of interest proportional to the total number of 16S rRNA gene copies per gram (g) of stool. For total bifidobacteria, only RA will be expressed.
Infant age at initial colonization with bacterial strains | Up to 60 days of age
  Age at initial colonization can only be defined at the level of the infant and will refer to each infant's first age (in days) at which colonization was detected or predicted to have occurred. This age may be derived empirically or using longitudinal modeling of infant-specific abundance trajectories. Colonization is a dichotomous variable that will be defined as an absolute abundance of a particular organism that exceeds a specified threshold. The term colonization refers here to the empirical detection of bacterial DNA at or above a particular level of abundance in stool, and will be used as a surrogate of intestinal colonization (in the absence of direct measurement of specific sites within the intestine).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roth, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Bangladesh (2):
  - Maternal Child Health Training Institute, Dhaka
  - Mohammadpur Fertility Services Training Centre, Dhaka